CLINICAL TRIAL: NCT02976792
Title: Effectiveness of the NephroCheck™ to Predict Postoperative Acute Kidney Injury in Patients Undergoing a Transcatheter Aortic Valve Implantation
Brief Title: Effectiveness of the NephroCheck™ After TAVI
Acronym: AKI-TAVI
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Principal Investigator, Alexandre OUATTARA, Head of department of Cardiovascular Anesthesia and Critical care, University Hospital, Bordeaux
Other Study IDs: DC 2016/94
Record Dates: First submitted 2016-10-11; First posted 2016-11-29 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Transcatheter Aortic Valve Implantation; Acute Kidney Injury; Postoperative Acute Renal Failure
Keywords: Transcatheter aortic valve implantation; Acute Kidney Injury; early acute kidney injury detection; Nephrocheck™; Renal Resistive Index
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Renal Resistive Index/NephroCheck™test: Patients undergoing a transcatheter aortic valve implantation
  Interventions: Procedure: Renal Resistive Index/NephroCheck™test

INTERVENTIONS:
Procedure: Renal Resistive Index/NephroCheck™test — Renal Resistive Index and NephroCheck™ test before TAVI and after TAVI

SUMMARY:
Postoperative acute renal failure is a frequent complication after a Transcatheter Aortic Valve Implantation (TAVI). The current practice cannot predict Acute Kidney Injuries (AKI) early enough to prevent an organic dysfunction triggering, consequently, cortical tubular necrosis.

Several recent studies in cardiac surgery have shown that sonographic criteria, the Renal Resistive Index (IRR), and a urinary biomarker, the NephroCheck™, could predict AKI promptly. These markers, sonographic and biologic, have both the advantage to be non-invasive and easy to perform. Each marker seems to have sensitivity and specificity to predict AKI promptly after cardiac surgery. Therefore, the IRR and the NephroCheck™ test could become essential tests to guide clinicians in determining rapidly whether a patient will develop AKI after a TAVI procedure. However, so far, no study has tested the NephroCheck™ in patients undergoing TAVI.

Therefore, the aim of this prospective observational study will be first to determine the effectiveness of the NephroCheck™ to predict AKI at an early stage after a TAVI procedure. The secondary outcome will be to compare the NephroCheck™ with the RRI in predicting at an earlier stage than the traditional method an AKI.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to undergo a TAVI

Exclusion Criteria:

* Chronic dialysis patients with anuria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a TAVI procedure
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the NephroCheck™ test to detect AKI after TAVI | Evolution of the Nephrocheck test from the time 0 to time 2.(Time 0: at inclusion before the TAVI / Time 1: NephroCheck™ Test at the first micturition post TAVI / Time 2: NephroCheck test™ on the first post operative day at the first micturition.)
  Determine the efficacy of NephroCheck™ test to predict AKI after TAVI. AKI will be defined according to the KADIGO criteria.

SECONDARY OUTCOMES:
Renal Resistive Index compared with NephroCheck™ | Evolution of the Renal Resistive Index from time 0 to time 2. Time 0: at inclusion before the TAVI / Time 1: at the first micturition post TAVI/ Time 2: on the first post operative day at the first micturition.
  compare the NephroCheck™ with the Renal Resistive Index in predicting an AKI

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre OUATTARA, MD, PhD, Principal Investigator — head of anesthesia department II
Locations (1):
- BORDEAUX UNIVERSITY HOSPITAL - Haut Lévêque, Pessac, France

IPD SHARING:
Plan to Share IPD: No